CLINICAL TRIAL: NCT04889521
Title: Impact of Distal Sensory Polyneuropathy on Function in Persons Living With HIV
Brief Title: Neuropathy Walks (Cross-sectional)
Status: Completed | Type: Observational
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, David Kietrys, Associate Professor, Rutgers, The State University of New Jersey
Other Study IDs: Pro2020003234(cross-sec)
Record Dates: First submitted 2021-05-11; First posted 2021-05-17 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: HIV Infections
Keywords: peripheral neuropathy; pain; function
MeSH Terms: conditions — HIV Infections; Peripheral Nervous System Diseases; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HIV and painful neuropathy: Persons living with HIV who also have painful distal sensory polyneuropathy in the feet.
  Interventions: Other: No intervention
- HIV without painful neuropathy: Persons living with HIV who do NOT have painful distal sensory polyneuropathy in the feet.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention. Study is cross-sectional observational.

SUMMARY:
Cross-sectional study is to explore the impact of painful neuropathy in the feet on function in persons living with HIV (PLHIV).

DETAILED DESCRIPTION:
The overall goal of this study is to explore the impact of HIV-associated distal sensory polyneuropathy on physical performance, physical activity, and pain pressure threshold.

The aim is to determine if the presence of painful distal sensory polyneuropathy in the feet adversely affects physical performance, physical activity, and pain pressure threshold in PLHIV.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of HIV infection currently treated with antiretroviral therapy (ART)
* cluster of differentiation 4 cell (CD4 cell) count of at least 200 cells/mm3
* 18-64 years of age
* able to read and write in English
* means to travel to a study site
* Additional inclusion for cohort with painful neuropathy in the feet:
* presence of peripheral neuropathy symptoms in feet
* average daily self-reported pain in the feet of at least 3/10 on a 0-10 numerical pain scale
* pain in the feet present for at least the past 3 months
* no changes in medications used to manage pain in the past 4 weeks

Exclusion Criteria:

* current opportunistic infection(s)
* cluster of differentiation 4 cell (CD4 cell) count <200 cells/mm3
* dementia
* uncontrolled psychiatric disorder
* wounds or sores on the feet
* musculoskeletal or neurological conditions (other than distal sensory neuropathy) that may affect gait
* pregnancy

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons living with HIV. Half of sample will include concurrent painful distal sensory neuropathy in the feet.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2024-09-13 (Actual); Study Completion 2024-09-13 (Actual)

PRIMARY OUTCOMES:
Gait - Walking velocity | Week 0 (one-time)
  Temporal characteristic of gait measured in m/sec as captured with a ZENO instrumented walkway
Gait - Step Length | Week 0 (one-time)
  Spatial characteristic of gait measured in meters as captured with a ZENO instrumented walkway
Gait - Step Time | Week 0 (one-time)
  Temporal characteristic of gait measure in seconds as captured with a ZENO instrumented walkway
Gait - Stride Width | Week 0 (one-time)
  Spatial characteristic of gait measured in meters as captured with a ZENO instrumented walkway
Gait - Cadence | Week 0 (one-time)
  Temporal characteristic of gait measured in steps per minute as captured with a ZENO instrumented walkway
Gait - Foot Fall Area | Week 0 (one-time)
  Spatial characteristic of gait measured in square meters as captured with a ZENO instrumented walkway
Physical Performance | Week 0 (one-time)
  Physical performance score generated via the Short Physical Performance Battery. (SPPB). SPPB procedures generate a total score reflective of physical performance. Minimum score=0; maximum score=12; lower score=worse outcome

SECONDARY OUTCOMES:
Walking Endurance | Week 0 (one-time)
  Walking endurance as measured with the 6-Minute Walk test (distance walked over span of 6 minutes).
Whole Body Strength | Week 0 (one-time)
  Mid-thigh pull test will be used to generate a score expressed as force in pounds or kilograms that is reflective of whole body strength.
Pain pressure threshold | Week 0 (one-time)
  Pain pressure threshold (expressed in pounds or kilograms of force) at lower extremity landmarks via use of a digital algometer
Physical Activity | 5 days from date of all other outcomes
  Physical activity characteristics: (1) over a span of 5 days captured via a wrist-band style Actigraph activity monitor; (2) self-reported physical activity over past 7 days using International Physical Activity Questionnaire - Short Form

CONTACTS AND LOCATIONS:
Overall Officials: David Kietrys, PhD, Principal Investigator — Rutgers School of Health Professions
Locations (2):
- United States (2):
  - Rutgers Physical Therapy Program, Blackwood, New Jersey
  - Rutgers Physical Therapy Program, Newark, New Jersey

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-18): https://cdn.clinicaltrials.gov/large-docs/21/NCT04889521/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-02): https://cdn.clinicaltrials.gov/large-docs/21/NCT04889521/ICF_001.pdf